CLINICAL TRIAL: NCT07404072
Title: Evaluation of Locally Applied Ferulic Acid as Adjunct to Mechanical Debridement in Treatment of Periodontitis (Clinical and Laboratory Study)
Brief Title: Evaluation of Locally Applied Ferulic Acid as Adjunct to Mechanical Debridement in Treatment of Periodontitis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Salah Awad Alanazi (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor-Investigator, Salah Awad Alanazi, B.D.S( Alfarabi University, 2019. Riyadh, KSA) Master Dgree at Oral Medicine, Periodontology, Diagnosis and Oral Radiology department (2021) Affiliation: Mansoura University, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ferulic acid in periodontitis
Record Dates: First submitted 2025-12-21; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis
Keywords: local drug delivery
MeSH Terms: conditions — Periodontitis | interventions — ferulic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ferulic Acid (Active Comparator): Drug Group
  Interventions: Drug: Ferulic Acid
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Scaling only (Other)
  Interventions: Procedure: mechanical debridement only
- Healthy (No Intervention)

INTERVENTIONS:
Drug: Ferulic Acid — Group 1: 20 Patients will be treated with Ferulic acid nanoparticles gel as an adjunct to mechanical debridement.
  Arms: Ferulic Acid
Drug: Placebo — 20 Patients will be treated with placebo gel as an adjunct to mechanical debridement
  Arms: Placebo
Procedure: mechanical debridement only — 20 Patients will be treated with mechanical debridement only
  Arms: Scaling only

SUMMARY:
to clinical evaluation of locally applied Ferulic acid nanoparticles as an adjunct to mechanical debridement in treatment of periodontitis

DETAILED DESCRIPTION:
Periodontitis is a complex chronic multifactorial inflammatory disease that impacts the tissues supporting teeth, causing their progressive destruction. It is initiated by bacterial infection, primarily involving Gram-negative anaerobic bacteria that trigger an immune response and production of pro-inflammatory cytokines. These cytokines recruit numerous neutrophils and macrophages to the site of infection resulting in the release of reactive oxygen species (ROS) and thus worsens tissue damage. Additionally, systemic diseases like diabetes mellitus or behaviors like smoking are examples of exacerbating factors .

Periodontitis remains a significant public health issue as it is the main cause of tooth loss and chewing dysfunction. This condition has far-reaching implications, affecting not only an individual's ability to maintain proper nutrition but also their quality of life and self-esteem. The impact of periodontitis extends beyond personal health, creating substantial socioeconomic burdens and escalating medical costs .

Therefore, effective treatment and management of periodontitis are crucial to mitigating these adverse effects and improving overall well-being. Tailored treatment approaches are essential, primarily focused on controlling the patient's infection. Supra- and subgingival instrumentation, commonly referred to as scaling and root planing (SRP), along with diligent home dental care, have an important role in managing the infection in patients diagnosed with periodontitis .

Systemic drugs used as adjuncts to SRP aim to enhance periodontal treatment outcomes by targeting bacterial pathogens or modulating the host immune response. Common systemic adjuncts include antibiotics, such as amoxicillin and metronidazole, which result in improvement in the clinical attachment levels (CAL) and reduction in periodontal probing depth (PPD) in chronic periodontitis patients. However, their prolonged use can lead to antibiotic resistance, gastrointestinal discomfort, and allergic reactions . Additionally, host-modulating agents, like sub-antimicrobial-dose doxycycline (SDD), inhibit matrix metalloproteinases (MMPs), reducing inflammation and tissue breakdown, but may cause photosensitivity or gastrointestinal issues with long-term use . Nonsteroidal anti-inflammatory drugs (NSAIDs) can also decrease bone resorption but are associated with gastrointestinal and cardiovascular side effects . While systemic drugs can augment SRP efficacy, their side effects and the potential for resistance necessitate careful patient selection and judicious use .

Optimizing the effectiveness of pharmacological therapy while minimizing risks and controlling the release of the drug is crucial. That's why a local drug delivery system (LDDS) is recommended in combination with SRP. LDDS shows promise in treating localized infections in various body parts and serves as a valuable tool for adjunctive local pharmacological therapy in periodontal treatment. LDDSs regulate the discharge of locally administered drugs meant to supplement periodontal treatment .

Ferulic acid, known as 4-hydroxy-3-methoxycinnamic acid, is a phenolic compound naturally found in various plants, including cereals, fruits, vegetables, and Chinese herbal medicines. It is known for its potent antioxidant properties, which help neutralize harmful free radicals and reduce oxidative stress. It also has numerous physiological properties, including anti-inflammatory, antioxidant, antibacterial, and anticancer, with low toxicity . In addition to being a free radical scavenger, ferulic acid also inhibits the enzymes that cause free radicals to form and increases the activity of scavenging enzymes . In addition, it is frequently used in skin care products as a brightening ingredient, photoprotective agent, and skin photoaging delayer .

Furthering, ferulic acid is one of the most important roles of phenolic acids, especially cinnamic acid derivatives, is their antioxidant activity, which depends primarily on the number of hydroxyl and methoxy groups attached to the phenyl ring. Ferulic acid is more easily absorbed into the body and stays in the blood longer than any other phenolic acids. Therefore, it is considered to be a superior antioxidant .

Hence, this study aimed to assess the validity of locally delivered ferulic acid nanoparticles as an adjunct to mechanical debridement for managing periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes 25-55 y.
* Patients who are systemically healthy,
* Patient exhibiting periodontal pocket depths (PD) ≥5mm,
* Presence of clinical attachment loss (CAL) between 3-4mm,
* Cooperative individuals capable of adhering to mechanical oral hygiene instructions

Exclusion Criteria:

* nPatients with sensitivity to the medication used in the study,
* Patients with a history of antibiotic use or anti-inflammatory drugs during the previous 3 months prior to the study,
* Patients with systemic diseases,
* Pregnant and lactating females,
* Smokers and tobacco chewers,
* Patients are not compliant with oral hygiene procedures.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in Probing Pocket Depth (PPD) | Baseline and 3 months after treatment
  Assessment of changes in probing pocket depth at selected periodontal sites to evaluate the clinical effectiveness of locally applied ferulic acid as an adjunct to mechanical debridement in patients with periodontitis.
Change in Clinical Attachment Loss (CAL) | Baseline and 3 months after treatment
  Evaluation of changes in clinical attachment loss to determine periodontal tissue response following adjunctive treatment with locally applied ferulic acid.

SECONDARY OUTCOMES:
Change in Gingival Index (GI) | Baseline and 3 months after treatment
  Measurement of gingival inflammation severity using the Gingival Index to assess the anti-inflammatory effect of locally applied ferulic acid.
Change in Plaque Index (PI) | Baseline and 3 months after treatment
  Assessment of dental plaque accumulation using the Plaque Index to evaluate changes in oral hygiene status following treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansura Universtiy, Al Mansurah, Mansura, Egypt

IPD SHARING:
Plan to Share IPD: Undecided